CLINICAL TRIAL: NCT06046027
Title: Efficacy of P6 Acupressure Band For Prevention of Postoperative Nausea and Vomiting In Children: A Randomized Controlled Trial
Brief Title: P6 Acupressure Band for Prevention of Postoperative Nausea and Vomiting in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FF-2019-413
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Nausea and Vomiting; Postoperative Nausea and Vomiting (PONV)Acuppressure
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accupressure Group (Experimental): Patient in Accupressure Group applied an acupressure band (ACU-STRAPTM) on bilateral hands with a plastic bead at P6 acupoint, which is situated at the wrist between the tendons of the palmaris longus and flexor carpi radialis, 2 cun proximal from the distal palmar crease as shown in Figure 1, half an hour prior to surgery at the operation theatre reception
  Interventions: Device: Accupressure band
- Placebo Group (Placebo Comparator): Patients in Placebo Group will receive a standard elastic band without acuppresure bead, which will be applied to the patient's wrist.
  Interventions: Device: Accupressure band

INTERVENTIONS:
Device: Accupressure band — The accupressure band and wirst band will be place 20 minutes prior to induction of anaesthesia. The induction and maintenance of anaesthesia performed at the discretion of the supervising anaesthesiologist. The maintenance of anaesthesia was achieved by administering sevoflurane at a minimum alveolar concentration (MAC) range of 1 to 1.2. A fresh gas flow rate of 2 L/min comprising a 50:50 concentration mixture of oxygen and air were employed. The patients will be ventilated and maintain end-tidal carbon dioxide (ETCO2) levels within the range of 35-40mmHg. All patients were administered intravenous dexamethasone at a dosage of 0.1mg/kg as a conventional prophylaxis for postoperative nausea and vomiting (PONV) following the induction of anaesthesia. Additionally, intravenous morphine was administered at a dosage of 0.05mg/kg and suppositories containing paracetamol were given at a dosage of 30mg/kg for analgesic purposes. Patients will be extubated at the end of surgery

SUMMARY:
Nausea and vomiting after surgery are one of the most common side effects of general anaesthesia. Pressure at P6 acupuncture point around wrist area using acupressure band has been proven to reduce nausea and vomiting in adult. We would like to see if this acupressure band can reduce nausea and vomiting in children after surgery.

Prior to operation, we will apply an elastic band at the P6 acupoint on your child's both hands. Your child will undergo anaesthesia as per usual and surgery as planned, with the elastic band onboard. Upon completion of surgery, your child will be required to wear the band and should not be removed. Your child will be monitored for up to 24 hours for episodes of nausea and vomiting. If so, rescue antivomit medication will be given. After 24 hours, we will record your level of satisfaction with the regimen provided

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) are the second most prevalent complaint among paediatric patients and is one of the most complex and serious concerns in anaesthetic practice. In addition to causing the patient misery and discomfort, nausea and vomiting can decrease parental satisfaction, increase the risk of pain and bleeding, increase resource utilisation, and lengthen the stay in the postoperative ward and hospital. In all paediatric populations, the incidence ranges from 13 to 42%, making it twice as prevalent as in adults[1].

The Eberhart categorization system for risk assessment of postoperative vomiting in paediatric patients encompasses several factors, namely age beyond 3 years, surgical length exceeding 30 minutes, undergoing strabismus surgery, and having a personal or family history of postoperative nausea and vomiting (PONV). The occurrence rates of postoperative nausea and vomiting (PONV) are reported as 10%, 20%, 50%, and 70% when one, two, three, or four risk factors are present, respectively [2]. A range of pharmacological and non-pharmacological approaches have been documented for the prevention and treatment of postoperative nausea and vomiting (PONV). Among the several non-pharmacological methods, acupoint stimulation appears to be the most promising approach[1].

The stimulation of acupoints can be classified as invasive and non-invasive techniques. Acupressure, a form of non-invasive acupoint stimulation, has been performed by the Chinese for over 2500 years[3]. It uses magnets, pellets, electrical stimulation, or micro beads to trigger the central nervous system, either locally or from a distance3. It is based on the idea that life energy moves through "meridians" in the body. When physical pressure is put on these meridians, it is meant to clear any blockages. Instead of using needles, acupressure includes putting pressure (usually with fingertips) on certain points on the body[3]. A Cochrane review and meta-analysis of the different ways to stimulate acupoints at the traditional Chinese Pericardium 6 (P6) point to avoid PONV shows that it works better than a placebo in adults[4, 5].

Research conducted on paediatric patients undergoing adenoidectomy or tonsillectomy has examined the efficacy of different acu-stimulation techniques, such as electroacupuncture and a combination of needle acupuncture and acupressure band, in comparison to standard care involving the use of dexamethasone. The findings of these studies indicate a statistically significant decrease in the occurrence of retching or vomiting among children who received acu-stimulation methods, as opposed to those who received standard care.[6, 7] In a systematic review conducted on a sample of 844 children, different approaches to administering acupoint stimulation at P6 were evaluated. The findings of this study revealed a statistically significant decrease in vomiting when compared to the control groups, which included Sham, placebo control, and conventional treatment.[8] This study postulates that the use of acupressure at the P6 acupoint in children, utilising an acupressure band, may provide an additional reduction in the occurrence of postoperative nausea and vomiting when combined with normal care. The objective of this study was to evaluate the efficacy of acupressure bands targeting the P6 acupoint in mitigating post-operative nausea and vomiting (PONV) among paediatric patients and to compare the postoperative need for metoclopramide between the group of patients using P6 acupressure bands and the group using a placebo.

ELIGIBILITY:
Inclusion Criteria:

* General surgery including open and laparoscopic hernia, orchidopexy surgery, orthopaedic and ENT surgery
* Duration of surgery of more than 30 mins and less than 4 hour
* ASA I or II

Exclusion Criteria:

* Inflammation over the relevant acupressure point and abnormal upper limb anatomy
* Planned admission to PACU/ICU post-operative or requiring mechanical ventilation post-operative
* Patient on antiemetic prior to surgery
* Known allergy to metoclopramide
* Suspected circulation or vascular problem of upper limb
* Upper limb surgery - strabismus surgery

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Incident of nausea and vomiting within 24 hours post operatively | up to 24 hours post surgery
  Incident of nausea and vomiting will be recorded in recovery area and hourly until 24H

SECONDARY OUTCOMES:
Numbers of rescue antiemetic needed | up to 24 hours post surgery
  Dosage and frequency of rescue antiemetic prescribed postoperatively will be recorded

OTHER OUTCOMES:
Complications | up to 24 hours post surgery
  Incident of complications related to accupressure band such as pain and redness
Parental satisfaction | up to 24 hours post surgery
  Degree of parental satisfaction by likert scale, 1 of very unsatisfied, 3 neutral and 5 very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon request

REFERENCES:
- [Background] Lee A, Chan SK, Fan LT. Stimulation of the wrist acupuncture point PC6 for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2015 Nov 2;2015(11):CD003281. doi: 10.1002/14651858.CD003281.pub4. PMID 26522652
- [Background] Chernyak GV, Sessler DI. Perioperative acupuncture and related techniques. Anesthesiology. 2005 May;102(5):1031-49; quiz 1077-8. doi: 10.1097/00000542-200505000-00024. PMID 15851892
- [Background] Eberhart LHJ, Geldner G, Kranke P, Morin AM, Schauffelen A, Treiber H, Wulf H. The development and validation of a risk score to predict the probability of postoperative vomiting in pediatric patients. Anesth Analg. 2004 Dec;99(6):1630-1637. doi: 10.1213/01.ANE.0000135639.57715.6C. PMID 15562045